CLINICAL TRIAL: NCT05350007
Title: Evaluation of Rumination, Frailty and Tanatophobia in Cancer Patients Over 65 Years of Age
Acronym: CANFRADE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Elif Yıldırım Ayaz, Principal Investigator, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: CANFRADE
Record Dates: First submitted 2022-04-18; First posted 2022-04-27 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Cancer; Death; Rumination; Frailty
Keywords: cancer; tanatophobia; rumination; fraility; elderly
MeSH Terms: conditions — Neoplasms; Death; Rumination Syndrome; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate tanatophobia and rumination in individuals over 65 years of age receiving cancer chemotherapy and to determine the related factors.

DETAILED DESCRIPTION:
No studies were found in the literature evaluating the relationship between frailty and lack of social support with tanatophobia and rumination. The aim of this study is to evaluate tanatophobia and rumination in individuals over 65 years of age receiving cancer chemotherapy and to determine the related factors.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* Conscious and no communication problems
* Being literate
* Willing to participate in our study voluntarily
* Cancer patient receiving active chemotherapy treatment

Exclusion Criteria:

* Not being willing to participate in the research
* Serious life-threatening condition (critical illness, intensive care unit stay, acute complication)
* Dementia, Alzheimer's, cognitive dysfunction
* Major psychiatric illness

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Cancer patients aged 65 and over receiving chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Rumination | 1 week
  Evaluation of rumination in patients over 65 years of age receiving cancer chemotherapy
Tanatophobia | 1 week
  Evaluation of tanatophobia in patients over 65 years of age receiving cancer chemotherapy

SECONDARY OUTCOMES:
fraility | 1 month
  Evaluation of fraility in patients over 65 years of age receiving cancer chemotherapy
lack of social support | 1 month
  Evaluation of lack of social support in patients over 65 years of age receiving cancer chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yıldırım Ayaz, M.D., Principal Investigator — Sultan Abdülhamid Training And Research Hospital
Locations (1):
- Sultan Abdülhamid Training and Research Hospital, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided